CLINICAL TRIAL: NCT05478135
Title: A Remote Evaluation of NAVIFY Oncology Hub Using Clinical Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prova Health Limited (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HLR-NOH-001
Record Dates: First submitted 2022-07-22; First posted 2022-07-28 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Oncology
Keywords: Digital Health; Health tech; Clinical simulation; Healthcare technology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NAVIFY Oncology Hub (Experimental): We will first conduct a small number of simulation sessions (3-5) to validate study methods and data collection procedures. Study methods may then be refined before conducting simulation sessions with a larger number of participants (approx. 25). In this phase, each participant will participate in a 90-minute simulation session in which they will use NAVIFY Oncology Hub to review synthetic patient cases. Participants will be tasked with reviewing the cases as if they were preparing to see a patient in a real clinical setting.
  Interventions: Device: NAVIFY Oncology Hub

INTERVENTIONS:
Device: NAVIFY Oncology Hub — NAVIFY Oncology Hub is a platform that aggregates and organizes disparate data into an intuitive, longitudinal view of the patient's cancer care journey. The platform is designed to optimize and support oncology workflows and decision-making by providing quick access to the most relevant data in one place, so that providers can make decisions more efficiently and collaborate more seamlessly.

SUMMARY:
This work seeks to understand current clinical workflow practice and validate use cases for NAVIFY Oncology Hub.

The main purpose of NAVIFY Oncology Hub is to enhance clinical and operational effectiveness, from diagnostic workup to treatment planning and management. This might free up providers' time and capacity to provide better and more personalized care to patients.

This research protocol builds on previous work that validated clinical simulation methods as a means for clinicians to generate useful insights during the testing and development of digital health tools (Gardner et al. 2020).

Accordingly, this study aims to test the ability of NAVIFY Oncology Hub to increase the work efficiency of oncologists and reduce the cognitive burden/mental fatigue associated with patient care and decision-making.

The insights generated will be used to guide the development of NAVIFY Oncology Hub and optimise user experience, as well as provide a better understanding of the opportunities for it to have maximal impact in the decision-making process.

DETAILED DESCRIPTION:
NAVIFY Oncology Hub is a platform that aggregates and organizes disparate data into an intuitive, longitudinal view of the patient's cancer care journey. The platform is designed to optimize and support oncology workflows and decision-making by providing quick access to the most relevant data in one place, so that providers can make decisions more efficiently and collaborate more seamlessly.

Clinical workflow is critical for the efficient and safe delivery of patient care. In most healthcare settings, clinical workflow is highly complex, and reflects the multidisciplinary collaboration and communication required of most clinical tasks. Studies have demonstrated a positive association between leveraging health information technology workflow tools for care coordination and patient engagement, and improved process quality metrics in preventive screening, diabetes control, as well as maternal and child health (Kruse & Bean 2018; Kranz et al. 2018). Embedded decision support tools have also been proven to improve the performance of risk assessments conducted by providers, as well as enhance patient safety and decrease mortality (Chaudhry et al. 2006; Wells et al. 2008; Jones et al. 2014; Campanella et al. 2015).

A set of 10 synthetic breast cancer patient cases will be developed by Prova Health. Cases will include history and examination findings, pathology reports, radiology reports and images (USS, mammogram, CT as applicable) and reports on tumor characteristics. The case details will be representative of a long term patient journey, inclusive of treatment lines such as adjuvant and neoadjuvant therapies. Cases will be selected to span the range of potential case scenarios seen in typical practice. Specifically, cases will be selected to include common invasive breast cancers (eg. IDC, ILC), as well as less common invasive breast cancers (eg. inflammatory). Cases will also represent a range of cancers with different molecular subtypes, such as whether the patient is HER2 positive or negative, hormone receptor (HR) positive or negative or triple negative. Finally, cases will also reflect the presentation of patients at various stages (eg. primary diagnosis, locally and regional advanced breast cancer, recurrent breast cancer, or metastatic advanced breast cancer).

Each participant will participate in a 90-minute remote (e.g., online) simulation session. During scheduling, participants will be given a link to use to join the session. This link will take them to a video conference call hosted through Google Meet. At the session, the moderator will facilitate the session and take notes.

Participants will use NAVIFY Oncology Hub to review synthetic patient cases. Participants will be tasked with reviewing the cases as if they were preparing to see a patient in a real clinical setting. This task will involve searching for, identifying, reviewing and synthesizing relevant clinical information (demographic information, pathology reports, clinical course, etc.) that supports decision-making. As such, this task is meant to simulate the same activities they would perform in their typical practice before inviting a patient into the clinic room for a consultation, and will permit this study to examine the usage of NAVIFY Oncology Hub on those activities.

Ultimately, the aim of the study is to investigate how NAVIFY Oncology Hub improves efficiency and reduces cognitive burden associated with reviewing and synthesizing patient information, and having participants engage with the platform requires them to go through those tasks.

ELIGIBILITY:
Inclusion Criteria:

* Board-certified, US-based oncologist
* Minimum 50% spent in clinical practice
* Active member of a tumor board

Exclusion criteria:

* Experience using NAVIFY Oncology Hub
* Inability to speak English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saira J Ghafur, MD, Principal Investigator — Prova Health Limited
Locations (1):
- Prova Health Limited, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This study will not share IPD

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27 US oncologists who are actively practicing and treat breast cancer were recruited during August and September 2022. Participants were affiliated with a healthcare institution where they are an active member of a tumor board and spend at least 50% of their time in clinical practice.
Period: Overall Study
Arm/Group | Navify Oncology Hub
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Navify Oncology Hub
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27
Board certification [Count of Participants; unit: Participants] — Board-certified US oncologists
  Participants | 27

OUTCOME MEASURES:

1. Primary Outcome: System Usability Scale (SUS)
Description: The System Usability Scale (SUS) a reliable tool for measuring the usability. It consists of a 10-item questionnaire with five response options for respondents; from Strongly disagree to Strongly agree. The participant's scores for each question added together and multiplied by 2.5 to convert the original scores of 0-100. A SUS score above a 68 would be considered above average and anything below 68 is below average.
Time Frame: 90 mins
Measure: Mean (95% Confidence Interval); unit: score on SUS
Arm/Group | Navify Oncology Hub
Number analyzed (Participants) | 27
score on SUS | 82 [75 to 89]

2. Primary Outcome: Participant-reported Efficiency When Preparing for Patient Consultations, Likert Scale
Description: Count of participants self-reporting that they were "a lot more efficient" or "somewhat more efficient" when using navify Oncology Hub to review patient information.
Time Frame: 90 mins
Measure: Count of Participants; unit: Participants
Arm/Group | Navify Oncology Hub
Number analyzed (Participants) | 27
Participants | 26

3. Primary Outcome: NASA Task Load Index (NASA-TLX)
Description: Number of participants who required "low" or "very low" levels of mental demand, temporal demand, and effort to successfully complete tasks using NAVIFY Oncology Hub.
Time Frame: 90 mins
Measure: Count of Participants; unit: Participants
Arm/Group | Navify Oncology Hub
Number analyzed (Participants) | 27
Participants | 17

4. Primary Outcome: Participant-reported Efficacy of Using Navify Oncology Hub to Facilitate Patient Discussions and Collaborate Care
Description: Number of participants self-reporting who felt nOH would be "significantly better" or "somewhat better" than their existing solution at facilitating patient discussion and coordinating care.
Time Frame: 90 mins
Measure: Count of Participants; unit: Participants
Arm/Group | Navify Oncology Hub
Number analyzed (Participants) | 27
Participants | 21

5. Primary Outcome: Participant-reported Fidelity of Synthetic Patient Cases
Description: Number of participants self-reporting that the synthetic patient cases were either 'very similar' or 'somewhat similar' to cases seen in routine clinical practice
Time Frame: 90 mins
Measure: Count of Participants; unit: Participants
Arm/Group | Navify Oncology Hub
Number analyzed (Participants) | 27
Participants | 25

ADVERSE EVENTS:
Time Frame: 3 hours
Description: 3 hours
Arm/Group | Navify Oncology Hub
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT05478135/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT05478135/ICF_001.pdf